CLINICAL TRIAL: NCT07013097
Title: A Single-center, Randomized, Double-blind, Placebo-controlled, Dose Escalation Phase I Clinical Study to Evaluate the Safety, Tolerability and Pharmacokinetics of PG-033 by Single Dose Administration and Food Effect in Healthy Volunteers
Brief Title: A Phase I Clinical Trial to Evaluate the Single Dose Ascending and Food Effects of PG-033 in Healthy Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Prime Gene Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PG-033-ND-101; CTR20251749 (Other: http://www.chinadrugtrials.org.cn/index.html)
Record Dates: First submitted 2025-05-19; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Lichen Simplex Chronicus
Keywords: PG-033; Lichen Simplex Chronicus; Pruritus
MeSH Terms: conditions — Neurodermatitis; Pruritus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Ascending Doses of PG-033 tablets (Active Comparator)
  Interventions: Drug: PG-033
- Placebo (Placebo Comparator)
  Interventions: Drug: PG-033 placebo comparator

INTERVENTIONS:
Drug: PG-033 — Oral tablets (2mg， 10mg)
  Arms: Single Ascending Doses of PG-033 tablets
Drug: PG-033 placebo comparator — Oral tablets (2 mg, 10 mg) (matching corresponding study medication)
  Arms: Placebo

SUMMARY:
The goal of this study is to evaluate the safety, tolerability and pharmacokinetics (PK) profiles of single ascending oral doses(SAD) of PG-033 by directly comparing it with placebo. Meanwhile, the impact of a high-fat meal on the pharmacokinetics of PG-033 will also be evaluated. The research will also explore the potential metabolites and metabolic pathways of PG-033 within the human body，as well as investigate the effect of PG-033 on the QTc interval.

DETAILED DESCRIPTION:
This is a single-center, randomized, double-blind, placebo-controlled, single-dose administration, and dose escalation phase I clinical study in adult participants aged from 18 to 45 years old (including threshold) with healthy male and female subjects. The study includs a single dose ascending study (SAD) and a food effect (FE) study.

The single ascending dose (SAD) study will be conducted by increasing the dosage from low dosage level to high. Approximately 40 participants will be randomized 3:1 to PG-033 or placebo in 5 dose groups.

The food effect study adopts a single-center, randomized, open-label, single-dose, two-period and two-sequence crossover clinical trial design. 12 participants will be randomly divided into group A and group B, with 6 participants in each group. In the first period, the 6 subjects in Group A will take PG-033 on an empty stomach, while the 6 subjects in Group B will take PG-033 after having a high-fat meal. In the second period, the two groups will cross over in taking the drug. That is, the subjects in Group A will take PG-033 after having a high-fat meal, and the subjects in Group B will take PG-033 on an empty stomach. The washout period between the two dosing periods is 7 days.

ELIGIBILITY:
Inclusion Criteria:

* 1. Read, understood, and signed an ICF before any investigational procedure(s) are performed.

  2.Male or female aged 18 to 45 (including threshold). 3. For male subjects, the body weight should be ≥ 50.0 kg, and for female subjects, the body weight should be ≥ 45.0 kg. The body mass index (BMI) should be within the range of 19.0 to 26.0 kg/m²(including threshold).

  4. Results of vital signs examination, physical examination, clinical laboratory tests (including blood routine examination, urine routine examination, blood biochemistry examination, coagulation function examination, thyroid function examination, etc.), chest X-ray, adrenal gland color ultrasound, etc. during the screening period show normal results or, if there are abnormalities, they are judged by the investigator to have no clinical significance.

  5. Be willing to avoid pregnancy or voluntarily take effective contraceptive measures and have no sperm or egg donation plan from the signing of the informed consent form to three month after the last administration of the investigational medicinal product.

  6. Be able to communicate well with the investigator and understand and comply with the requirements of the study.

Exclusion Criteria:

* 1. Participants with abnormal electrocardiogram results during screening (e.g., QT/QTcF > 440 ms, PR interval > 200 ms, QRS complex duration > 100 ms, clinically significant abnormalities of the P wave, clinically significant changes in the ST-T wave, etc.).

  2. Participants known to be allergic to this product or related excipients; or participants with an allergic constitution (such as those who are allergic to two or more drugs or foods).

  3. Participants with a history of chronic diseases or severe diseases in the circulatory, urinary, respiratory, hematological and lymphatic, endocrine, immune, mental and neurological, digestive systems, etc.

  4. Participants who have undergone major surgery within 6 months before the first dose administration, or those who plan to have surgery during the study period, or those who have undergone surgery that, as judged by the investigator, will affect the evaluation of the drug's safety and pharmacokinetic characteristics.

  5. Participants who have used any drugs (including any prescription drugs, over-the-counter drugs, traditional Chinese herbal medicines) and health products within 2 weeks before the first dose administration.

  6. Participants who have used any drugs that inhibit or induce the liver's metabolism of drugs (e.g., barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole, selective serotonin reuptake inhibitors (SSRI) antidepressants, cimetidine, diltiazem, macrolides, nitroimidazoles, sedative-hypnotics, verapamil, fluoroquinolones, antihistamines, etc.) within 4 weeks before the first dose administration.

  7. Participants who are unable to stop consuming beverages and foods containing caffeine, alcohol, etc. (including chocolate, tea, coffee, cola, etc.), or foods that affect drug metabolism such as grapefruit, grapefruit products, pitaya, mango, pomelo, etc. from 48 hours before the first dose administration until the end of the trial, or those who are unable to stop consuming the above-mentioned diets from 48 hours before the first dose administration until the end of the trial.

  8. Participants who have received live attenuated vaccine vaccination within 4 weeks before the first dose administration or those who need to receive live attenuated vaccine vaccination during the trial.

  9. Participants with positive serological results for hepatitis B surface antigen (HBsAg), hepatitis C antibody, Treponema pallidum antibody, or human immunodeficiency virus antibody during screening.

  10. Participants who have participated in other clinical trials within 3 months before the first dose administration.

  11. Participants who have donated blood or lost a total of ≥ 400 mL of blood (excluding physiological blood loss in females) within 3 months before the first dose administration, received blood transfusion or used blood products, or those who plan to donate blood during the trial or within 1 month (30 days) after the end of the trial.

  12. Participants who have consumed an average of more than 2 units of alcohol per day within 30 days before screening (1 unit ≈ 360 mL of beer or 45 mL of liquor with an alcohol content of 40% or 150 mL of wine), or those who cannot abstain from alcohol during the trial, or those with a positive result in the alcohol breath test.

  13. Participants who have smoked an average of more than 5 cigarettes per day within 3 months before screening, or those who cannot stop smoking during the trial.

  14. Participants with a history of drug abuse within 1 year before screening or those who tested positive for drug abuse screening.

  15. Participants who cannot tolerate intravenous puncture/indwelling needle or those with a history of fainting at the sight of needles or blood.

  16. Participants with special dietary requirements and who cannot accept the unified diet.

  17. Pregnant or lactating women; 18. Other participants determined by the investigator to be unsuitable for participation.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-05-23 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of PG-033 tablets | Single Ascending Dose study: 7 days；Food Effect study: 14 days
  Incidence of treatment-emergent adverse events (AEs) and serious adverse events (SAEs)

SECONDARY OUTCOMES:
Pharmacokinetics parameter: Cmax | up to 3 days
  Maximum Observed Plasma concentration (Cmax)
Pharmacokinetics Parameter:Tmax | up to 3 days
  Time at which the maximum plasma concentration (Cmax) occurs
Pharmacokinetics parameter: AUC0-t | up to 3 days
  Area under the plasma concentration-time curve from dosing (time zero） to the time of the last measured concentration
Pharmacokinetics parameter: AUC0-∞ | up to 3 days
  Area Under the Plasma Concentration Versus Time Curve from Zero Extrapolated to Infinity (AUC0-∞）
Pharmacokinetics parameter: t1/2 | up to 3 days
  Terminal Elimination Half-Life (t1/2)
Pharmacokinetics parameter: Vd/F | up to 3 days
  Volume of Distribution (Vd/F)
Pharmacokinetics parameter: CL/F | up to 3 days
  Total Body Clearance
Pharmacokinetics parameter: λZ | up to 3 days
  Elimination rate constant (λz)
Pharmacokinetics parameter: MRT | up to 3 days
  Mean retention time (MRT)
Corrected QT interval | up to 24 hours post-dose
  Change in QT interval corrected for heart rate (QTc) interval from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Shijitan Hospital , Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No